CLINICAL TRIAL: NCT04776746
Title: An Open-Label Extension Study of Continuing Treatment With Trofinetide for Rett Syndrome
Brief Title: Open-Label Extension Study of Trofinetide for Rett Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: As a result of marketing approval of trofinetide on 10 March 2023, the study was terminated by the Sponsor with the intent of switching patients to commercially available product.
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-2566-005
Record Dates: First submitted 2020-11-29; First posted 2021-03-02 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome | interventions — trofinetide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug - trofinetide (Experimental): trofinetide oral solution
  Interventions: Drug: trofinetide

INTERVENTIONS:
Drug: trofinetide — Study drug is administered twice a day for up to approximately 32 months. Doses may be taken orally or administered by gastrostomy (G) tube. The subject's assigned dose for this study will be the final dose from the antecedent study (ACP-2566-004).

SUMMARY:
To investigate the safety and tolerability of continued long-term treatment with oral trofinetide in girls and women with Rett syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Has completed the EOT visit of the antecedent trofinetide Study ACP-2566-004 (i.e., has completed 40 weeks)
2. May benefit from continued treatment with open-label trofinetide in the judgment of the Investigator
3. Can still swallow the study medication provided as a liquid solution or can take it by gastrostomy tube
4. The subject's caregiver is English-speaking and has sufficient language skills to complete the caregiver assessments

   Childbearing Potential
5. Subjects of childbearing potential must abstain from sexual activity for the duration of the study and for at least 30 days thereafter. If a subject is sexually active or becomes sexually active during the study, she must use 2 clinically acceptable methods of contraception (e.g., oral, intrauterine device [IUD], diaphragm plus spermicide, injectable, transdermal or implantable contraception) for the duration of the study and for at least 30 days thereafter. Subject must not be pregnant or breastfeeding.

Exclusion Criteria:

1. Began treatment with growth hormone during the antecedent study
2. Began treatment with IGF-1 during the antecedent study
3. Began treatment with insulin during the antecedent study
4. Has developed a clinically significant cardiovascular, endocrine (such as hypo- or hyperthyroidism, Type 1 diabetes mellitus, or uncontrolled Type 2 diabetes mellitus), renal, hepatic, respiratory, or gastrointestinal disease (such as celiac disease or inflammatory bowel disease)
5. Subject is judged by the Investigator or the Medical Monitor to be inappropriate for the study due to AEs, medical condition, or noncompliance with investigational product or study procedures in the antecedent study
6. Has a clinically significant abnormality in vital signs at Baseline
7. Has an average QTcF interval of >450 ms on the Baseline ECG performed before the first dose of trofinetide is given in the present study (i.e., the ECG performed at the EOT visit of the antecedent study)
8. Has developed a clinically significant ECG finding during the antecedent study

Additional inclusion/exclusion criteria apply. Patients will be evaluated at baseline to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically, if it is determined that their baseline health and condition do not meet all pre-specified entry criteria).

Ages: 5 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 77 (Actual)
Dates: Start 2020-11-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Translational Genomics Research Institute (TGen), Phoenix, Arizona
  - University of California, San Diego, La Jolla, California
  - UC Davis MIND Institute, Sacramento, California
  - Children's Hospital Colorado Aurora, Aurora, Colorado
  - University of South Florida, Tampa, Florida
  - Emory Genetics Clinical Trial Center, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Kennedy Krieger Institute, John Hopkins School of Medicine, Baltimore, Maryland
  - Boston Children's Hospital Harvard Medical School, Boston, Massachusetts
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Greenwood Genetic Center, Greenwood, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Percy AK, Neul JL, Benke TA, Berry-Kravis EM, Glaze DG, Marsh ED, Barrett AM, An D, Bishop KM, Youakim JM. Trofinetide for the treatment of Rett syndrome: Long-term safety and efficacy results of the 32-month, open-label LILAC-2 study. Med. 2024 Oct 11;5(10):1275-1281.e2. doi: 10.1016/j.medj.2024.06.007. Epub 2024 Jul 17. PMID 39025065
- [Derived] Parent H, Ferranti A, Niswender C. Trofinetide: a pioneering treatment for Rett syndrome. Trends Pharmacol Sci. 2023 Oct;44(10):740-741. doi: 10.1016/j.tips.2023.06.008. Epub 2023 Jul 16. PMID 37460385

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, open-label, long-term study of trofinetide to monitor the safety and efficacy of continuing trofinetide therapy for patients who previously completed a Phase 3 trofinetide study. Patients who completed the preceding open-label study ACP-2566-004 were eligible to enroll in this study. Study ACP-2566-004 was an extension study for randomized, double-blind, placebo-controlled study ACP-2566-003.
Groups:
- Trofinetide: Trofinetide oral solution was administered twice daily for a planned duration of up to approximately 32 months, orally or administered by gastrostomy (G) tube. Treatment duration could be less than 32 months if trofinetide became commercially available during the study, or if development of trofinetide for Rett syndrome was discontinued.
Period: Overall Study
Arm/Group | Trofinetide
Started | 77
Completed | 0
Not Completed | 77
Not completed — Study terminated by sponsor | 61
Not completed — Adverse Event | 5
Not completed — Death | 4
Not completed — Lack of Efficacy | 3
Not completed — Noncompliance with study drug | 2
Not completed — Not related to COVID-19 | 2

BASELINE CHARACTERISTICS:
Population: All patients enrolled and treated with trofinetide
Groups:
- Trofinetide: Trofinetide oral solution was administered twice daily for up to approximately 32 months, orally or administered by gastrostomy (G) tube. The patient's assigned dose for this study was the final dose from the antecedent study (ACP-2566-004).
Arm/Group | Trofinetide
Number analyzed (Participants) | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.0 (4.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 71
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 77

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Treatment-emergent Adverse Events (TEAEs), With Serious Adverse Events (SAEs), and With Withdrawals Due to AEs
Description: Withdrawals due to AEs included both study drug discontinuation as well as study termination
Time Frame: Mean study drug exposure was 426 days, corresponding to 1.2 years
Population: All patients enrolled and treated
Measure: Count of Participants; unit: Participants
Arm/Group | Trofinetide
Number analyzed (Participants) | 77
Participants
  Patients with TEAEs | 68
  Patients with SAEs | 23
  Patients with AEs leading to discontinuation | 9

2. Primary Outcome: Number (%) of Patients With Potentially Clinically Important Changes in ECG Post-baseline
Description: Potentially clinically significant ECG changes were defined as QTcF >500 ms or QTcF change from baseline (CFB) of >60 ms
Time Frame: Mean study drug exposure was 426 days, corresponding to 1.2 years
Population: All patients enrolled and treated
Measure: Count of Participants; unit: Participants
Arm/Group | Trofinetide
Number analyzed (Participants) | 77
Participants
  QTcF >500 ms | 0
  QTcF CFB >60 ms | 1

3. Primary Outcome: Number (%) of Patients With Potentially Clinically Important Changes in Vital Signs Post-baseline
Description: Potentially clinically important changes from baseline in vital signs were defined as:
  Systolic blood pressure (SBP) ≥180 mmHg and increased ≥20 mmHg from baseline; SBP ≤90 mmHg and decreased ≥20 mmHg from baseline; Diastolic blood pressure (DBP) ≥105 mmHg and increased ≥15 mmHg from baseline; DBP ≤50 mmHg and decreased ≥15 mmHg from baseline; Pulse rate (PR) ≥120 bpm and increased ≥15 bpm from baseline; PR≤50 bpm and decreased ≥15 bpm from baseline. Baseline was the baseline value of previous study ACP-2566-003.
Time Frame: Mean study drug exposure was 426 days, corresponding to 1.2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Trofinetide
Number analyzed (Participants) | 77
Participants
  SBP≥180 mmHg and increased ≥20 mmHg from BL | 0
  SBP≤90 mmHg and decreased ≥20 mmHg from BL | 5
  DBP≥105 mmHg and increased ≥15 mmHg from BL | 1
  DBP≤50 mmHg and decreased ≥15 mmHg from BL | 4
  PR≥120 bpm and increased ≥15 bpm from BL | 4
  PR≤50 bpm and decreased ≥15 bpm from BL | 0

4. Primary Outcome: Number (%) of Patients With Potentially Clinically Important Changes in Body Weight Post-baseline
Description: Potentially clinically important changes from baseline in body weight were defined as:
  Weight increase ≥7% from baseline Weight decrease ≥7% from baseline
Time Frame: Mean study drug exposure was 426 days, corresponding to 1.2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Trofinetide
Number analyzed (Participants) | 77
Participants
  Weight increase ≥7% from BL | 45
  Weight decrease ≥7% from BL | 9

5. Primary Outcome: Number (%) of Patients With Potentially Clinically Important Changes in Laboratory Parameters Post-baseline
Description: Potentially clinically important changes in laboratory parameters were defined as: sodium ≤125 mmol/L; sodium ≥155 mmol/L; potassium ≤3.0 mmol/L ; potassium ≥5.5 mmol/L; chloride ≤85 mmol/L; chloride ≥120 mmol/L; calcium <2.0 mmol/L; calcium >2.75 mmol/L; blood urea nitrogen ≥10.71 mmol/L; creatinine >1.5× upper limit of normal (ULN); uric acid ≥505.75 μmol/L; lactate dehydrogenase (LDH) ≥3×ULN; glucose ≤2.48 mmol/L; glucose ≥11 mmol/L; albumin ≤26 g/L; albumin ≥60 g/L; protein ≤50 g/L; protein ≥100 g/L; alanine transaminase (ALT) ≥3×ULN; aspartate transaminase (AST) ≥3×ULN; gamma glutamyl transferase (GGT) ≥3×ULN; alkaline phosphatase (ALP) ≥3×ULN; bilirubin ≥1.5×ULN
Time Frame: Mean study drug exposure was 426 days, corresponding to 1.2 years
Population: All patients enrolled and treated and with at least one postbaseline value for the respective parameter (n=75; apart from deviating patient numbers of n=74 for uric acid, LDH, AST and bilirubin)
Measure: Count of Participants; unit: Participants
Arm/Group | Trofinetide
Number analyzed (Participants) | 75
Participants
  Sodium ≤125 mmol/L | 0
  Sodium ≥155 mmol/L | 0
  Potassium ≤3.0 mmol/L | 1
  Potassium ≥5.5 mmol/L | 0
  Chloride ≤85 mmol/L | 0
  Chloride ≥120 mmol/L | 0
  Calcium <2.0 mmol/L | 0
  Calcium >2.75 mmol/L | 0
  Blood urea nitrogen ≥10.71 mmol/L | 0
  Creatinine >1.5× ULN | 0
  Uric acid ≥505.75 μmol/L: number analyzed (Participants) | 74
  Uric acid ≥505.75 μmol/L | 0
  LDH ≥3×ULN: number analyzed (Participants) | 74
  LDH ≥3×ULN | 0
  Glucose ≤2.48 mmol/L | 1
  Glucose ≥11 mmol/L | 1
  Albumin ≤26 g/L | 0
  Albumin ≥60 g/L | 0
  Protein ≤50 g/L | 0
  Protein ≥100 g/L | 0
  ALT ≥3×ULN | 2
  AST ≥3×ULN: number analyzed (Participants) | 74
  AST ≥3×ULN | 0
  GGT ≥3×ULN | 2
  ALP ≥3×ULN | 1
  Bilirubin ≥1.5×ULN: number analyzed (Participants) | 74
  Bilirubin ≥1.5×ULN | 0

ADVERSE EVENTS:
Time Frame: Mean study drug exposure was 426 days, corresponding to 1.2 years
Arm/Group | Trofinetide
All-Cause Mortality (participants affected / at risk) | 4/77
Serious Adverse Events (participants affected / at risk) | 23/77
Other Adverse Events (participants affected / at risk) | 57/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trofinetide (N=77)
Cardiac arrest (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Sudden unexplained death in epilepsy (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (4)
COVID-19 (Infections and infestations) | 1 (1)
Enterovirus infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Renal procedural complication (Injury, poisoning and procedural complications) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Seizure (Nervous system disorders) | 5 (6)
Disturbance in attention (Nervous system disorders) | 1 (1)
Dystonia (Nervous system disorders) | 1 (1)
Dystonic tremor (Nervous system disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Pelvic fluid collection (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trofinetide (N=77)
Diarrhoea (Gastrointestinal disorders) | 13 (18)
Vomiting (Gastrointestinal disorders) | 10 (12)
Constipation (Gastrointestinal disorders) | 9 (9)
Pyrexia (General disorders) | 12 (20)
COVID-19 (Infections and infestations) | 20 (22)
Urinary tract infection (Infections and infestations) | 12 (21)
Upper respiratory tract infection (Infections and infestations) | 9 (13)
Influenza (Infections and infestations) | 6 (6)
Pharyngitis streptococcal (Infections and infestations) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 4 (4)
Pneumonia (Infections and infestations) | 4 (5)
Viral upper respiratory tract infection (Infections and infestations) | 4 (4)
Electrocardiogram QT prolonged (Investigations) | 4 (4)
Weight decreased (Investigations) | 4 (4)
Seizure (Nervous system disorders) | 8 (11)
Lethargy (Nervous system disorders) | 4 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5)

LIMITATIONS AND CAVEATS:
As a result of marketing approval of trofinetide on 10 March 2023, the study was terminated by the Sponsor with the intent of switching patients to commercially available product. Date of study termination was 30 June 2023.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to his/her own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT04776746/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT04776746/SAP_001.pdf